CLINICAL TRIAL: NCT05148273
Title: Investigation of the Effects of Telehealth Applications Applied to Infertile Women During Drug Treatment Procedures on Anxiety Levels: A Randomized Controlled Study
Brief Title: The Effect of Telehealth Applications on the Level of Anxiety in the Treatment of Infertility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Basak Demiralp Yavuz, principal investigator, Suleyman Demirel University
Other Study IDs: TELENURSING and anxıety
Record Dates: First submitted 2021-11-04; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Infertility
Keywords: Infertility; telehealth; anxiety; consultancy
MeSH Terms: conditions — Infertility; Anxiety Disorders | interventions — Telenursing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intervention: After the selection process with 1 to 1 randomization method, a personal information form and Beck anxiety scale will be applied to the women selected for the case group on the day of the initiation of treatment with assisted reproductive techniques interview. Then, within an average of 10 days, there is a treatment procedure including planned drug use, messages containing drug doses, drug use, drug administration, follicle count, reminder of the times of operations such as OPU, IUI, ET, and motivational issues. Medication use, time, date, dose, application form and motivational sentences will be sent every day through the WhatsApp application. The Beck anxiety scale will be repeated on the day of IUI and ET procedures, and the effect of telehealth practices on the anxiety levels of women undergoing infertility treatment will be evaluated. During the study, the participants will be able to reach the researcher from their mobile phones whenever they want.
  Interventions: Behavioral: telenursing
- control: In the first interview at the beginning of the treatment protocol with assisted reproductive techniques, a personal information questionnaire and beck anxiety scale will be applied to the control group selected by the 1-to-1 randomization method. Afterwards, the Beck anxiety scale will be applied again at the end of the treatment without any intervention.

INTERVENTIONS:
Behavioral: telenursing — 7-24 counseling and daily treatment protocol reminders will be given to the intervention group.
  Groups: intervention

SUMMARY:
It is expected that 84% natural pregnancy will occur at the end of the first 12 months of sexual intercourse without the use of contraceptive methods.The lack of natural fertility is under the influence of multiple factors. These factors can be summarized as age, past infections, genetic factors, anatomical structural disorders, environmental toxins, occupational exposure, lifestyle and sexually transmitted infections.Severe psychological stress, anxiety and depression are encountered in the diagnosis, treatment method and management of the related process in couples who are faced with the diagnosis of infertility.

With the telehealth service that came to the fore in the world in the 1950s, nurses use it in the management of many treatment processes such as infertility treatment, with the roles of managing the information collection process, making decisions with the information they receive, and transmitting information on patients who are far away and need constant follow-up.

Assisted reproductive technologies, which are the current treatment method of infertility, have been used effectively for thirty years. Anxiety control is important in the success of treatment in the treatment process, which is both costly and stressful. Providing 24/7 hours of counseling by using telehealth methods contributes to the reduction of this anxiety.

DETAILED DESCRIPTION:
Ethics committee and hospital approval were obtained in order to conduct the study. The sample of the study consists of people who applied to the IVF clinic of Süleyman Demirel University Research and Practice Hospital. The work is planned to be completed between April 2021 and March 2022. In the first meeting with the participants, it is carried out by taking precautions to protect against the COVID 19 pandemic, in cases where it is met face to face. Participants will be divided into groups with 1 to 1 method in randomization. Participants assigned to the intervention group will be given a personal information form and beck anxiety scale before treatment, followed by telehealth service throughout the treatment protocol, and the beck anxiety scale will be repeated at the end of the treatment. In the control group, a personal information form and Beck anxiety scale will be applied before the treatment and will be repeated after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 20-45
* Female
* Having been diagnosed with infertility
* Should be able to use a smart phone
* Open to communication

Exclusion Criteria:

* Not between the ages of 20-45
* Individuals who do not want to be inherited

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As a gender, it should carry the phenomena of the female gender anatomically and psychologically.
Study Population: The study consists of infertile women between the ages of 20-45 who applied to the in vitro fertilization clinic of the Süleyman Demirel University Research and Application Hospital in Isparta, Turkey.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
beck anxiety scale | 1 year
  The intervention group will be evaluated with the Beck anxiety scale at the beginning of the treatment. Afterwards, the patient who was given telehealth service throughout the treatment will be compared by applying the Beck anxiety scale again at the end of the treatment.
  The control group will be compared by applying the Beck anxiety scale before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: başak demiralp yavuz, nurse, Principal Investigator — researcher
Locations (1):
- Suleyman Demırel Unıversıty research and practice hospital, Isparta, Center, East Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since it is an ongoing thesis work, I do not want to share the data for a while.